CLINICAL TRIAL: NCT02448251
Title: A Phase I, Multicenter, Open-Label Safety, Pharmacokinetic and Preliminary Efficacy Study of Wild-type Sparing EGFR Inhibitor, AC0010MA, in Adult Patients With Previously Treated EGFRmut and Acquired T790M Mutation Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Safety, Pharmacokinetic and Preliminary Efficacy Study of AC0010MA in Advanced Non Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: ACEA Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC00102014-101
Record Dates: First submitted 2015-05-12; First posted 2015-05-19 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — abivertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- single dose per day (QD) (Experimental): Phase I Arm 1: AC0010MA orally taking once daily, starting from 100 mg per day.
  Interventions: Drug: AC0010MA
- two doses per day (BID) (Experimental): Phase I Arm 2: AC0010MA orally taking twice daily, starting from 200 mg per day (100 mg BID). Arm 2 will be initiated once the drug plasma t1/2 is 10 hours or below in the first dose cohort (100 mg QD).
  Interventions: Drug: AC0010MA

INTERVENTIONS:
Drug: AC0010MA — Following Phase I, a protocol amendment will be submitted to the IND to specify the selected dose and dose justification to be used in Phase II.

SUMMARY:
AC0010MA is a new, irreversible, Epidermal Growth Factor Receptor (EGFR) mutation selective Tyrosine Kinase Inhibitor. Aim at local advanced or metastatic non-small cell lung cancer patients with EGFR mutation or T790M drug-resistant mutation. The molecular mechanism: by irreversible combining the EGFR-RTKs ATP binding site of cell, selectively suppress the activities of EGFR tyrosine kinase phosphorylation, block the signal transduction pathway of EGFR and inhibit the function of ras/raf/MAPK downstream, thus block the tumor cell growth by EGFR induction, and promotes apoptosis. AC0010MA Maleate Capsules has three characters: 1. Irreversible binding to EGFR; 2. Effectively suppresses the tumor cell with EGFR mutant while has no suppression to EGFR wild-type cell; 3. Efficient suppress the tumor cell with EGFR T790M drug-resistant mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female, aged 18 years or older at the time of consent; preferably non-Asian.
2. Has histologically or cytologically confirmed metastatic, or unresectable locally advanced, recurrent NSCLC.
3. Has at least one measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI), according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
4. Has documented evidence of an activating EGFR mutation in the tumor tissue determined by either sequencing or PCR-based technique (Part 1).
5. For Part 1 only: subjects with a positive T790M mutation are preferred, but not required. Confirmation of T790M mutation status will be determined from an archived tumor tissue sample or fresh tumor tissue sample obtained via biopsy if archived tissue is not available. In Part 2, subjects must have a confirmed, positive T790M EGFR mutation (acquired T790M EGFR mutation or "de novo" T790M EGFR mutation).
6. Has a life expectancy of at least 3 months.
7. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Has adequate hematological and physiological functions.
9. Has documented disease progression while receiving at least 30 days of treatment with a currently approved EGFR tyrosine kinase inhibitor (TKI) (e.g., erlotinib, gefitinib or afatinib) with intervening treatment after most recent EGFR TKI therapy (not required for "de novo" T790M EGFR mutation).
10. Signed and dated written informed consent obtained prior to any study-specific evaluation.

Exclusion Criteria:

1. Has a history of interstitial lung disease related to prior EGFR inhibitor therapy.
2. Has an EGFR TKI- related toxicity that has NOT resolved to Grade 1 or less.
3. Is test positive for hepatitis C virus (HCV), hepatitis B virus (HBV) or human immunodeficiency virus (HIV) antibody.
4. Has received the prohibited therapy (e.g., concurrent anti-cancer therapy including but not limited to: chemotherapy, radiation, hormonal, or immunotherapy) ≤14 days prior to first planned dose of AC0010MA.
5. Received prior treatment with AZD9291 (osimertinib) or CO1686 (rociletinib) and experienced disease progression.
6. Is a female subject who is pregnant or breastfeeding.
7. Female subjects (if of child bearing potential) and male subjects (with a partner of child bearing potential) must use medically acceptable methods of birth control before study entry, for the duration of the study, and for at least 6 months after the last intake of study drug.
8. Has a serious or unstable concomitant systemic disorder incompatible with the clinical study (e.g., substance abuse, uncontrolled psychiatric condition, uncontrolled intercurrent illness including active infection, arterial thrombosis, or symptomatic pulmonary embolism).
9. Has any other reason(s) for the investigator to consider that the subject should not participate in the study.
10. Is receiving treatment with medication(s) that are known to be strong inhibitors or inducers of CYP3A4/5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability, and the maximum tolerated dose (MTD) of AC0010MA determined by incidence of dose limiting toxicity (DLT) | Within the first 28 days of treatment.
  To determine the safety and tolerability and to establish the maximum tolerated dose (MTD) of AC0010MA by incidence of dose limiting toxicity (DLT), defined as Grade 3 or 4 adverse events (AEs) and clinical lab abnormalities occurring within the first 28 days of treatment.

SECONDARY OUTCOMES:
Evaluation of tumor response and duration of response of AC0010MA ((objective response rate, ORR) | within the time frame of every 8 weeks (2 cycles) for up to 3 years
  To characterize tumor response (objective response rate, ORR) and duration of response of AC0010MA as a criterion for further development of AC0010MA in this patient population.
Maximum plasma concentration (Cmax) of AC0010MA | Blood samples will be collected at pre-treatment, and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 24h post-treatment on Days 1, 8, and 28 in the first treatment cycle (QD and BID) in Phase I
  To evaluate pharmacokinetic parameter of AC0010MA
Time to Cmax | Blood samples will be collected at pre-treatment, and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 24h post-treatment on Days 1, 8, and 28 in the first treatment cycle (QD and BID) in Phase I
  To evaluate pharmacokinetic parameter of AC0010MA
Terminal half-life (t1/2) | Blood samples will be collected at pre-treatment, and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 24h post-treatment on Days 1, 8, and 28 in the first treatment cycle (QD and BID) in Phase I
  To evaluate pharmacokinetic parameter of AC0010MA
Area under the plasma concentration-time curve | Blood samples will be collected at pre-treatment, and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 24h post-treatment on Days 1, 8, and 28 in the first treatment cycle (QD and BID) in Phase I
  To evaluate pharmacokinetic parameter of AC0010MA
Volume of distribution (V/F) | Blood samples will be collected at pre-treatment, and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 24h post-treatment on Days 1, 8, and 28 in the first treatment cycle (QD and BID) in Phase I
  To evaluate pharmacokinetic parameter of AC0010MA
Plasma Concentration (CL/F) | Blood samples will be collected at pre-treatment, and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 24h post-treatment on Days 1, 8, and 28 in the first treatment cycle (QD and BID) in Phase I
  To evaluate pharmacokinetic parameter of AC0010MA

CONTACTS AND LOCATIONS:
Overall Officials: Vali A. Papadimitrakopoulou, MD, Study Director — MD Anderson Cancer Center, Houston, TX, USA; Suresh S. Ramalingam, MD, Principal Investigator — Emory University School of Medicine, Atlanta, GA, USA; Heather Wakelee, MD, Principal Investigator — Stanford University, Palo Alto, CA, USA; Karen L Reckamp, MD, Principal Investigator — City of Hope Comprehensive Cancer Center, Duarte, CA, USA
Locations (8):
- United States (4):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Stanford University, Palo Alto, California
  - Emory University School of Medicine, Atlanta, Georgia
  - MD Anderson Cancer Center, Houston, Texas
- CEPCM - Hopital Timone, Marseille, France
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - START-Madrid-FJD, Madrid
  - START-Madrid-CIOCC, Madrid

IPD SHARING:
Plan to Share IPD: No